CLINICAL TRIAL: NCT05179096
Title: Randomized Trial on the Effects of a Mindfulness Intervention on Temperament, Anxiety and Depression: a Multi-arm Psychometric Study
Brief Title: Effects of a Mindfulness Intervention on Temperament, Anxiety and Depression: the Mind the Child Study
Acronym: MTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Andrea Poli, Dr., University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MTC-01
Record Dates: First submitted 2021-12-07; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Child, Only; Temperament; Anxiety; Depression
Keywords: Child; Mindfulness; Temperament; Anxiety; Depression; Attention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Participants in the experimental group will undergo an 8-week mindfulness training program with weekly 60-minute group sessions
  Interventions: Behavioral: Mindfulness-based intervention
- Control (No Intervention): The control group will follow routine daily school activities

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — The program consists of a series of awareness practices: the exercises are presented in progression, starting from the awareness of the external environment, then the self-awareness in the environment, the awareness of the body and the five senses, the awareness of the interconnection among the various forms of life and, eventually, meditation exercises that characterize the awareness of the cognitive processes
  Arms: Mindfulness

SUMMARY:
Background and study aims:

Mindfulness is a mental state that can be achieved through meditation. So far, studies have shown that practicing mindfulness on a consistent and regular basis can improve attentional functions and emotional well-being. Mindfulness has recently begun to be used in the field of child development. The aim of this study is to assess if a mindfulness program may help primary school students in reducing anxiety and depression while also improving their temperament.

Who can participate? Students attending the fourth or fifth year of primary school

What does the study involve? Participants will be randomly assigned to the experimental and control groups. Participants in the experimental group will undergo an 8-week mindfulness training program with weekly 60-minute group sessions, while the control group will follow routine daily school activities.

Questionnaires will be used to assess temperament, anxiety and depression before and after the intervention.

What are the possible benefits and risks of participating? Benefits of participating in the study may include a lowering of anxiety and depression levels, as well as an improvement of temperament.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 9 to 11 years
2. Children have reasonable comprehension of spoken language and can follow simple instructions
3. Children and their parents are willing to attend all intervention sessions
4. Children and parents have an adequate understanding of English

Exclusion Criteria:

1. Concurrent enrollment in other intervention trials
2. Child or parent regularly practice complementary health interventions such as meditation

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Temperament - Inhibition to Novelty (IN) | QUIT-IN is measured before and after the 8-week mindfulness intervention
  IN dimension of temperament is measured using Italian Questionnaires of Temperament (QUIT). Higher scores mean a worse outcome
Temperament - Attention (AT) | QUIT-AT is measured before and after the 8-week mindfulness intervention
  AT dimension of temperament is measured using Italian Questionnaires of Temperament (QUIT). Higher scores mean a better outcome
Temperament - Motor Activity (MA) | QUIT-MA is measured before and after the 8-week mindfulness intervention
  MA dimension of temperament is measured using Italian Questionnaires of Temperament (QUIT). No overall change is expected in MA scores
Temperament - Social Orientation (SO) | QUIT-SO is measured before and after the 8-week mindfulness intervention
  SO dimension of temperament is measured using Italian Questionnaires of Temperament (QUIT). Higher scores mean a better outcome
Temperament - Positive Emotionality (PE) | QUIT-PE is measured before and after the 8-week mindfulness intervention
  PE dimension of temperament is measured using Italian Questionnaires of Temperament (QUIT). Higher scores mean a better outcome
Temperament - Negative Emotionality (NE) | QUIT-NE is measured before and after the 8-week mindfulness intervention
  NE dimension of temperament is measured using Italian Questionnaires of Temperament (QUIT). Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Anxiety | TAD for Anxiety is measured before and after the 8-week mindfulness intervention
  Anxiety is measured using Anxiety and Depression Test in Childhood and Adolescence (TAD). Higher scores mean a worse outcome
Depression | TAD for Depression is measured before and after the 8-week mindfulness intervention
  Depression is measured using Anxiety and Depression Test in Childhood and Adolescence (TAD). Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Poli, Psy.D., Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
Raw data are available on request.
Supporting Information: Study Protocol